CLINICAL TRIAL: NCT05581888
Title: Visual Performance of Different Types of Functional Intraocular Lenses in Cataract Patients
Brief Title: Visual Performance of Functional Intraocular Lenses in Cataracts
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Functional IOLs in cataracts
Record Dates: First submitted 2022-09-19; First posted 2022-10-17 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: High Myopia; Cataract
Keywords: Visual performance; Trifocal IOL; High myopic cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 839MP group (Other): Patients in this group were binocularly implanted with the AT LISA tri 839MP trifocal intraocular lens.
  Interventions: Device: trifocal intraocular lens
- TFNT00 group (Other): Patients in this group were binocularly implanted with the AcrySof IQ PanOptix TFNT00 trifocal intraocular lens.
  Interventions: Device: trifocal intraocular lens

INTERVENTIONS:
Device: trifocal intraocular lens — Binocular implantation of two different trifocal intraocular lens in high myopic cataracts

SUMMARY:
This is a prospective, multi-center, randomized comparative study. The purpose of the study is to evaluate and compare the postoperative visual outcomes and quality of vision of two diffractive trifocal intraocular lenses (IOLs) in patients with high myopic cataracts.

DETAILED DESCRIPTION:
Binocular implantation of two types of trifocal IOLs was performed in patients with high myopic cataracts. Postoperative uncorrected distance (UNVA), intermediate (UIVA), near (UNVA), and best-corrected distance visual acuity (BCVA) were measured. Defocus curve, high-order aberrations, modulation transfer function curve, Strehl ratio and reading ability were compared between the two groups. The functional vision and incidence of photic phenomena were surveyed using questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* required binocular cataract extraction
* age > 21 years
* length of optic axis > 26 mm

Exclusion Criteria:

* irregular corneal astigmatism > 0.3 um;
* amblyopia; previous ocular surgery;
* ocular pathologies such as diabetic retinopathy, macular degeneration, glaucoma with field defects;
* requirements for further ocular surgery (other than Nd:YAG capsulotomy) or retinal laser treatments during the study

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
uncorrected distance visual acuity (UDVA) | one year
  uncorrected visual acuity at 5 m
best corrected distance visual acuity (BCVA) | one year
  corrected visual acuity at 5 m
uncorrected near visual acuity (UNVA) | one year
  uncorrected visual acuity at 40 cm
uncorrected intermediate visual acuity (UIVA) | one year
  uncorrected visual acuity at 60 cm

SECONDARY OUTCOMES:
HOAs | three months
  high order aberrations such as coma
Strehl Ratio | three months
  The derivative of point spread function (PSF)
objective visual quality | three months
  MTF curves

CONTACTS AND LOCATIONS:
Overall Officials: Jin Yang, Study Director — Department of Ophthalmology, Eye and Ear, Nose, and Throat Hospital, Fudan University
Locations (1):
- Eye & ENT Hospital of Fudan University, Shanghai, Shanghai Municipality, China